CLINICAL TRIAL: NCT06809348
Title: Development of PRECISE: a Data Driven Personalized Suicide Prevention Intervention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Kevin Kuehn, Assistant Adjunct Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 811796
Record Dates: First submitted 2025-01-24; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Suicidal Thoughts and Behaviors
Keywords: personalized interventions; intensive longitudinal data; emotion regulation; coping; coping skills; dialectical behavior therapy; cognitive behavior therapy; ecological momentary assessment; personalized feedback; technology; coaching
MeSH Terms: conditions — Suicidal Ideation; Behavior; Emotional Regulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-Intensity (Experimental): In the high intensity arm, participants will complete all eight weeks of EMA with idiographic models generated between each session. Coaches then shape selection of skills in collaboration with the patient and a treatment plan for the next session will be generated.
  Interventions: Behavioral: PRECISE
- Low-Intensity (Experimental): In the low intensity arm, participants will complete only an initial two weeks burst of EMA and GIMME will be run following an initial burst. A treatment plan for the next eight weeks will be generated based on the output.
  Interventions: Behavioral: PRECISE

INTERVENTIONS:
Behavioral: PRECISE — PRECISE includes aspects of several evidence-based approaches, such as Safety Planning and DBT to manage and reduce suicide risk. During the initial visit, staff train participants how to complete EMAs. Participants then complete two weeks of five-times per day EMAs regarding their emotions, emotion regulation strategies as well as SITBs. Following an initial "learning period", participant data is analyzed via GIMME to determine the within-person correlates of SITBs. Data is processed through a real-time pre-programmed data cleaning and analysis script. Coaches then teach a selection of skills in collaboration with the client.

SUMMARY:
Individuals at high-risk of suicide vary substantially from one another. Over time, risk factors for suicide may change within the same individual. Despite these differences, most treatments for suicidal thoughts assume that the same intervention works equally well for all individuals at high-risk of suicide. Intensive longitudinal data combined with network science, integrated with coaching, could be used to personalize suicide prevention interventions to make them more effective and efficient. This K23 Career Development application involves refining and testing a novel personalized treatment for individuals at high-risk called PeRsonalizEd Clinical Intervention for Suicidal Events or PRECISE. PRECISE leverages idiographic statistical techniques adopted from network science applied to ecological momentary assessment data to inform the tailoring of Safety Planning and skills from Dialectical Behavior Therapy, two existing evidence-based treatments for suicide. In Aim 1, a user-centered design approach will be used to refine PRECISE. Following the refinement of the intervention, informed by data from a case series in Aim 1, the investigators will then conduct a randomized controlled trial comparing two different intensities of personalization. In the low-intensity arm, the 8-week treatment will be tailored based on an initial two-week burst of ecological momentary assessment and one idiographic model. In the high-intensity arm, participants complete eight weeks of ecological momentary assessment and idiographic models are generated between each session. Coaches use the idiographic models to identify an individuals' drivers of suicidal thoughts and conduct behavioral chain analyses to tailor specific skills to then teach, shape, and reinforce in their individual clients. Assessments are completed pre-treatment, 8-weeks post-enrollment, and 16-weeks enrollment. The investigators hypothesize that both arms will demonstrate clinically significant reductions in suicidal ideation, but the high-intensity arm will be superior to the low-intensity arm in reducing ideation. Furthermore, the investigators anticipate that increases in effective emotion regulation skills and reductions in negative affect will account for the decrease in suicidal ideation. As individuals learn more effective emotion regulation strategies, they will experience less distress and thereby lower levels of suicidal ideation. This project is responsive to Objective 3.2 of the NIMH Strategic Plan and is integrated with a mentored research training plan focused on 1) suicide specific rigorous clinical trials, 2) user centered design in digital health, and 3) applications of network science to intensive longitudinal data. The project and training goal will support the Candidate's overarching goal to become a clinician-scientist engaged in independent research on personalized, impactful, rapid acting suicide prevention interventions for at risk adults.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Endorsement of active suicidal ideation on the Columbia Suicide Severity Rating Scale (>2 or past month thoughts of killing self or attempt in past month)
* English fluency
* Willingness to provide contact information for a key information to be contacted as part of our risk and safety plan.

Exclusion Criteria:

* Past year exposure to DBT
* Moderate/severe substance use disorder within the past thirty days
* Dementia, mild cognitive impairment and/or traumatic brain injury
* Lack of capacity to consent to research and/or under conservatorship.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Scale for Suicide Ideation | From enrollment to the end of the follow-up assessment at 6-months.
  The Beck Scale for Suicide Ideation (SSI) is a 21-item self-report scale that measure the intensity of suicidal thoughts. The MSSI ranges from 0 [min] to 63 [max] with higher scores suggesting more severe suicidal ideation.

SECONDARY OUTCOMES:
Emotion Reactivity Scale | From enrollment to the end of the follow-up assessment at 6-months.
  The ERS is a 21-item self-report measure developed to measure an individuals' emotion reactivity. The ERS ranges from 0 [min] to 84 [max] with higher scores suggesting more emotional intensity.
Cognitive Emotion Regulation Questionnaire | From enrollment to the end of the follow-up assessment at 6-months.
  The Cognitive Emotion Regulation Questionnaire (CERQ) is a 36-item, self-report, multidimensional questionnaire constructed in order to identify the cognitive emotion regulation strategies (or cognitive coping strategies) someone uses after having experienced negative events or situations. Participants rate the 36 items using a 5-point Likert style scale (1 = Almost Never; 2 = Sometimes; 3 = Frequently; 4 = Often; 5 = Almost Always). There are 9 sub scales of the CERQ; 1) self-blame 2) acceptance; 3) rumination; 4) positive refocusing; 5) refocus planning; 6) positive reappraisal; 7) putting things into perspective; 8) catastrophizing; and 9) blaming others. Sub scales are calculated by summing across the items and dividing by the number of items within each sub scale (4). Higher scores indicate more frequent use of the strategy.

CONTACTS AND LOCATIONS:
Locations (1):
- 8980 Villa La Jolla Drive, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The study data manager will ensure all data is uploaded to the NIMH National Data Archive in accordance with existing guidelines and upload timelines (also see Resource Sharing). Anonymous data may also be uploaded to public repositories (e.g., Open Science Framework, Github) to facilitate data sharing with other researchers and ensure accuracy in reporting results.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be uploaded to the Open Science Framework by 03/31/2030 and will be shared indefinitely.